CLINICAL TRIAL: NCT05926921
Title: 'The Effect of Musical Intervention on the Indicators of Pain in Newborns Undergoing IV-line Placement'
Brief Title: Musical Intervention During IV-line Placement in Neonates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaarne Gasthuis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: newwave
Record Dates: First submitted 2023-06-09; First posted 2023-07-03 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Pain
Keywords: intravenous line; newborn; music; pain management; musical therapy
MeSH Terms: conditions — Pain; Agnosia | interventions — Music Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music (Active Comparator): Brahms lullaby at 50-60dB (depending on distance to speaker), played during the intravenous line procedure.
  Interventions: Other: music
- no music (No Intervention): No intervention, care as usual.

INTERVENTIONS:
Other: music — Brahms' Lullaby will be played from a speaker at 50 decibels
  Arms: music

SUMMARY:
The goal of this clinical trial is to test the effect of music in reducing the pain felt by newborn children during an intravenous line procedure. An intravenous line is a small tube brought into a vein by using a needle. The main questions it aims to answer are:

1. Does playing a lullaby during intravenous line procedures affect the vital signs and behavior of a newborn, compared to not playing music?
2. How do parents and medical staff experience the music that's being played? Participants will all receive the same care and treatments as usual. The only difference being about half of the participants will be randomly assigned to the group that gets music.

Researchers will compare the music group to the non-music group to see if there is any difference in vital signs and behaviors of the child.

DETAILED DESCRIPTION:
After inclusion, a participant will be randomized by drawing a sealed, opaque envelope, the contents of which will be either group A: no music, or group B: music. The outcome assessor will then perform a baseline measurement of vital signs and Neonatal Infant Pain Score. Then, Brahms Lullaby will be played from a speaker. When the needle is first introduced into the skin, a second measurement will be performed. For every attempt needed to succesfully place the intravenous line, an additional measurement will be done. Finally, after succesful placement of the intravenous line is confirmed by NaCl flush, a final measurement will be done. Afterwards, a short questionnaire will be filled in by the parents and the medical staffmember(s) that performed the intravenous line.

The study groups will be compared to each other in outcome measures, and there will be statistical correction for demographic and clinical confounders, which will be collected from medical files. The research hypothesis is that group B will show a smaller increase in vital signs and NIPS on average during the procedure, compared to group A.

ELIGIBILITY:
Inclusion Criteria:

* connected to a monitor that records vital signs
* receives an IV-line

Exclusion Criteria:

* has hearing impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-10-09 (Estimated); Study Completion 2024-10-09 (Estimated)

PRIMARY OUTCOMES:
HR | one day
  heart rate
RR / BR | one day
  respiratory rate / breathing rate
O2 Sat | one day
  oxygen saturation
NIPS | one day
  neonatal infant pain scale

SECONDARY OUTCOMES:
parents' experience (questionnaire) | one day
  four short questions regarding parents' thoughts about the intervention
IV-line performers' experience (questionnaire) | one day
  four short questions regarding staff' thoughts about the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Spaarne Gasthuis Haarlem Zuid, Haarlem, North Holland, Netherlands